CLINICAL TRIAL: NCT02864615
Title: A Phase 1b Study of Safety and Preliminary Efficacy of Stereotactic Body Radiation Therapy (SBRT) in Patients With Metastatic Renal Cell Carcinoma Treated With Targeted or Immuno- Therapy (Volga Study).
Brief Title: Safety and Preliminary Efficacy of SBRT in Patients With Metastatic RCC Treated With Targeted or IO Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCRB29022016
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: renal cell carcinoma; metastasis; stereotactic body radiation therapy; targted therapy; immune checkpoint inhibitors
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Body Radiation Therapy (Experimental): Patients with stable disease on targeted or IO therapy will receive SBRT on first metastasis of clear cell renal cell carcinoma. Second metastasis will be as a control. In case of safety and 50% reduction in size of first metastasis, up to 10 metastasis will be treated with SBRT.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Dose and schedule will be depended on metastases location.

SUMMARY:
Aim of this phase 1b study is to evaluate safety and preliminary efficacy of stereotactic body radiation therapy in patients with metastatic renal cell carcinoma treated with VEGFR, mTOR or immune checkpoint inhibitors.

DETAILED DESCRIPTION:
This is prospective phase 1b study.

Patients with metastatic RCC receiving targeted or IO therapy (VEGFR inhibitor or mTOR inhibitor or checkpoint inhibitors in approved treatment lines and in standard therapeutic regimens) with stable diseaseor durable partial response for at least 4 months, are enrolled in the study.

The initial examination includes CT with contrast, where the selected measured 2 metastatic sites, stable for at least 4 months but no more than 6 months of targeted therapy (increase or decrease in size in the course of targeted therapy should not exceed 10%). Metastases have to be located in one organ. Allowed location of metastases: lungs, liver, lymph nodes, contralateral kidney, adrenal gland.

Size of selected metastases should not be less than 5 mm and not more than 4 cm.

ELIGIBILITY:
Inclusion Criteria:

1. clear cell renal cell carcinoma
2. confirmed distant metastases
3. previous nephrectomy
4. stable disease or durable partial response on recommended targeted and IO therapy
5. age: > 18 years
6. signed informed consent

Exclusion Criteria:

1. unability to select first and second metastases
2. history of serious cardiac arrhythmia, congestive heart failure, angina pectoris, or other severe cardiovascular disease (i.e., New York Heart Association class III or IV)
3. other malignancy
4. grade 3 and 4 toxicity of targeted therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events of SBRT | 4 months

SECONDARY OUTCOMES:
Rate of reduction in size of first metastasis exposed to radiation | 4 months
Time to progression of first (study) and second (control) metastases | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Tsimafeyeu, M.D., Study Director — Kidney Cancer Research Bureau; Natalia Dengina, M.D., Principal Investigator — Ulyanovsk Regional Cancer Center
Locations (1):
- Ulyanovsk regional cancer center, Ulyanovsk, Ulyanovsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dengina N, Mitin T, Gamayunov S, Safina S, Kreinina Y, Tsimafeyeu I. Stereotactic body radiation therapy in combination with systemic therapy for metastatic renal cell carcinoma: a prospective multicentre study. ESMO Open. 2019 Oct 13;4(5):e000535. doi: 10.1136/esmoopen-2019-000535. eCollection 2019. PMID 31673426